CLINICAL TRIAL: NCT04877249
Title: Gait Training to Reduce Compensatory Walking Patterns in Post-Stroke Hemiparesis
Brief Title: Gait Training in Post-Stroke Hemiparesis Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0091
Record Dates: First submitted 2021-04-07; First posted 2021-05-07 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Hemiparesis; Split-belt treadmill; gait training
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait training for stroke (Experimental)
  Interventions: Behavioral: Split-belt treadmill training
- Gait training for healthy (Active Comparator)
  Interventions: Behavioral: Split-belt treadmill training

INTERVENTIONS:
Behavioral: Split-belt treadmill training — 1. Split-belt gait training without or with any resistance, 2. Facilitating the knee extension during the terminal swing phase of gait cycle to identify the impact on the propulsive force generation of paretic leg

SUMMARY:
The focus of this study is to optimize the delivery of a combined strength and aerobic training regimen to individuals with post stroke hemiparesis and reduce overuse and inefficiencies associated with the nonparetic leg during walking. This study proposes to use 1) split-belt treadmill and 2) single belt treadmill walking using split belt simulation software for enhancing symmetrical walking patterns for people with stroke.

DETAILED DESCRIPTION:
This study will include twenty stroke survivors and twenty healthy adults (total 40 participants) who are 20 years or older. Both groups (stroke vs healthy) will be screened and recruited from a UTMB Stroke Support Group and local community in Galveston or Harris County for one year (2021-22). Healthy individuals will also participate in gait training compared to stroke participants. The focus of this gait training is to optimize the delivery of a combined strength and aerobic training regimen to older adults with post stroke hemiparesis and reduce overuse and inefficiencies associated with the nonparetic leg during walking. Investigators propose to use a combination of neuromechanical and biobehavioral approaches to enhance bilateral symmetry of limb propulsion using specialized split-belt, force-plate instrumented treadmill that uses backward directed resistance forces. With neuromechanics investigators will measure joint torque output, EMG muscle activity patterns, and trailing limb angle, while a person is walking under normal treadmill belt conditions versus the split-belt conditions at different levels of resistance. Electromyography (EMG) detects electrical activity during muscle contraction while the single or the split-belt treadmill walking. The joint torque output and trailing limb angle can be obtained by using the Vicon Motion System (Vicon, Oxford, UK) in conjunction with the Bertec split-belt, force plates instrumented treadmill (Bertec Corp., Columbus, OH). In addition, in terms of biobehavioral metrics, investigators will measure the extent to which people maintain improved paretic limb propulsion contributions immediately after the split-belt environment is restored to a single belt condition (i.e. aftereffects), and the ability of individuals to consciously alter their walking pattern so as to reduce compensatory walking patterns when they are not engaged with the specialized treadmill setup.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, ages 20 or older
* Healthy participants will be required to be medically stable
* Healthy participants are able to walk at least 10 meters independently at a comfortable speed without an assistive device
* The participants with a history stroke, ages 20 or older
* Unilateral first stroke of ischemic origin in the carotid artery distribution
* Unilateral first stroke of hemorrhagic origin in the carotid artery distribution
* Diagnosis of stroke at least 6 months prior to participation
* Free of major post-stroke complications (e.g., recurrent stroke, hip fracture, myocardial infarction)
* Living within the community
* The participants with a history stroke are able to ambulate 10 meters with or without assistive devices

Exclusion Criteria:

* A history of any significant orthopedic problems
* A history of psychiatric or cognitive illness (e.g., bipolar affective disorder, psychosis, schizophrenia, attention deficits, cognitive deficits, or medication refractor depression)
* Neurological problems
* Stroke secondary to subarachnoid hemorrhage or posterior circulation stroke
* Not expected to live more than one year
* Comatose
* Unable to follow 3 step commands
* Amputation
* Poorly controlled diabetes (e.g., foot ulceration)
* Blind
* Progressive neurological diseases
* Comprehensive aphasia
* Medical instability
* Significant musculoskeletal problems
* Congestive cardiac failure
* Unstable angina
* Peripheral vascular disease
* Neuropsychiatric disorders (e.g., dementia, cognitive deficits, and severe depression)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Bilateral symmetry of ground reaction forces during split-belt treadmill walking | Single point of assessment in one day and ground reaction forces will be recorded continuously for 20-30minutes and will be expressed per gait cycle
  Vertical, horizontal, and mediolateral ground reaction force changes will be measured in response to split/tied belt speed and with (or without) a resistance using the Bertec split-belt, force plates instrumented treadmill and the Vicon 3D motion analysis system.
Bilateral symmetry of joint torques during split-belt treadmill walking | Single point of assessment in one day and joint torques will be recorded continuously for 20-30minutes and will be expressed per gait cycle
  Joint torques changes of ankle, knee, and hip joints will be measured in response to split/tied belt speed and with (or without) a resistance using the Bertec split-belt, force plates instrumented treadmill and the Vicon 3D motion analysis system.
Trailing limb angle during split-belt treadmill walking | Single point of assessment in one day and trailing limb angle will be recorded continuously for 20-30minutes and will be expressed per gait cycle
  Peak trailing limb angle changes will be measured in response to split/tied belt speed and with (or without) a resistance using the Bertec split-belt, force plates instrumented treadmill and the Vicon 3D motion analysis system.
Bilateral muscles activities during split-belt treadmill walking | Single point of assessment in one day and muscle activity will be recorded continuously for 20-30minutes and will be expressed per gait cycle
  Timing (milliseconds) of Soleus, Tibialis Anterior, and Quadriceps muscle activities changes will be recorded continuously in response to split/tied belt speed and with (or without) a resistance using Delsys wireless EMG system.
Bilateral muscles activities during split-belt treadmill walking | Single point of assessment in one day and muscle activity will be recorded continuously for 20-30minutes and will be expressed per gait cycle
  Peak amplitude (millivolts) of Soleus, Tibialis Anterior, and Quadriceps muscle activities changes will be recorded continuously in response to split/tied belt speed and with (or without) a resistance using Delsys wireless EMG system.
Spatiotemporal patterns during split-belt treadmill walking | Single point of assessment in one day and spatiotemporal gait parameters will be recorded continuously for 20-30minutes and will be expressed per gait cycle.
  Cadence (Step numbers/minute) during split/tied treadmill walking will be recorded continuously using the Vicon 3D motion analysis system.
Spatiotemporal patterns during split-belt treadmill walking | Single point of assessment in one day and spatiotemporal gait parameters will be recorded continuously for 20-30minutes and will be expressed per gait cycle.
  Step and stride length (cm) during split/tied treadmill walking will be recorded continuously using the Vicon 3D motion analysis system.
Spatiotemporal patterns during split-belt treadmill walking | Single point of assessment in one day and spatiotemporal gait parameters will be recorded continuously for 20-30minutes and will be expressed per gait cycle.
  Stance and swing time (sec) during split/tied treadmill walking will be recorded continuously using the Vicon 3D motion analysis system.

SECONDARY OUTCOMES:
Spatiotemporal patterns of overground walking | Baseline assessment before split/tied treadmill walking
  Walking speed (m/sec) during overground walking will be recorded continuously using the Zeno Walkway system.
Spatiotemporal patterns of overground walking | Baseline assessment before split/tied treadmill walking
  Cadence (Step numbers/minute) during overground walking will be recorded continuously using the Zeno Walkway system.
Spatiotemporal patterns of overground walking | Baseline assessment before split/tied treadmill walking
  Step and stride length (cm) during overground walking will be recorded continuously using the Zeno Walkway system.
Spatiotemporal patterns of overground walking | Baseline assessment before split/tied treadmill walking
  Stance and swing time (sec) during overground walking will be recorded continuously using the Zeno Walkway system.
Kinematic representation of the temporal events during standing and walking | Baseline assessment before split/tied treadmill walking
  The temporal events of foot position (sec) will be identified from ground reaction forces (GRFs) during standing and walking trials using the Tekscan High Resolution Mat.
Kinematic representation of the temporal events during standing and walking | Baseline assessment before split/tied treadmill walking
  The standing balance (cm2) will be measured using sway analysis from Tekscan High Resolution Mat.

CONTACTS AND LOCATIONS:
Overall Officials: Mansoo Ko, Ph.D., Principal Investigator — University of Texas
Locations (1):
- School of Health Profession, University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moradian N, Ko M, Hurt CP, Brown DA. Effects of backward-directed resistance on propulsive force generation during split-belt treadmill walking in non-impaired individuals. Front Hum Neurosci. 2023 Dec 4;17:1214967. doi: 10.3389/fnhum.2023.1214967. eCollection 2023. PMID 38111676